CLINICAL TRIAL: NCT06858254
Title: Standard Optimization of Autologous Stem Cells by Intranasal and Intravenous Administration to Treat Parkinson's Disease and Atypical Parkinsonism
Brief Title: Standard Optimization of Stem Cells in Parkinson's Disease and Atypical Parkinsonism
Acronym: SO-ASC-INIVAT
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Apeiron Research Center (Other)
Collaborators: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Jason Glowney, Principal Investigator/Medical Director, Apeiron Research Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ARC-PD-PPS-01
Record Dates: First submitted 2025-02-19; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Atypical Parkinsonism; Parkinson Disease (PD)
Keywords: Atypical Parkinsonism; Parkinson-Plus Syndrome; Stem Cells; MSCs; Epigenetics; Metagenomics; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Parkinson Disease Group 1 (Experimental): Day 0 - Sham IV + INA BMAC 6 months - IV BMA + Sham INA 12 months - IV BMA + INA BMAC
  Interventions: Biological: Autologous mesenchymal stem cells
- Parkinson Plus Syndrome Group 1 (Experimental): Day 0 - Sham IV + INA BMAC 6 months - IV BMA + Sham INA 12 months - IV BMA + INA BMAC
  Interventions: Biological: Autologous mesenchymal stem cells
- Parkinson Disease Group 2 (Experimental): Day 0 - IV BMA + Sham INA 6 months - Sham IV + INA BMAC 12 months - IV BMA + INA BMAC
  Interventions: Biological: Autologous mesenchymal stem cells
- Parkinson Plus Syndrome Group 2 (Experimental): Day 0 - IV BMA + Sham INA 6 months - Sham IV + INA BMAC 12 months - IV BMA + INA BMAC
  Interventions: Biological: Autologous mesenchymal stem cells

INTERVENTIONS:
Biological: Autologous mesenchymal stem cells — 1. Participant's blood is drawn at the start of each visit.
  2. Bone marrow aspirate is drawn from the posterior aspect of the pelvis and is subsequently harvested and processed.
  3. The following procedures are administered in a crossover design (Day 0 and 6 months):
     * Intranasal bone marrow aspirate administration (INA BMAC) OR Sham INA
     * Intravenous bone marrow aspirate administration (IV BMA) OR Sham IVA
  4. At 12 months, all participants receive IV BMA + INA BMAC

SUMMARY:
The purpose of this study is to measure outcomes using intranasal and intravenous autologous bone marrow mesenchymal stem cells (BM-MSCs) for Parkinson Disease (PD) and Parkinson's Plus (PPS) patients.

DETAILED DESCRIPTION:
Parkinson Disease (PD) and Parkinson-Plus Syndrome (PPS) are complex neurodegenerative diseases (NDDs) affecting more than 10 million people worldwide. The clinical application of stem cell therapy holds great promise in the treatment of NDDs by promoting regeneration and modulating immune responses with bone marrow aspirate, in particular, holding considerable potential in neural repair and recovery. However, current approaches often rely on university-based laboratories and invasive delivery approaches, raising patient safety, accessibility, and cost concerns. Additionally, NDDs present with distributive and heterogenous pathology, complicating treatment strategies. As pharmaceutical and biotech companies develop targeted stem cell therapies, most focus on localized brain structures rather than targeting PD/PPS systemically. Advancing consensus between scientific research and clinical application is critical for earlier detection in the prodromal phase, identifying epigenetic risk factors, and developing therapeutics that provide a broader, more effective treatment.

The primary objective of this study is to measure outcomes using autologus bone marrow mesenchymal stem cells (BM-MSCs) on motor and non-motor function in persons with PD/PPS. The trial will include 60 participants (40 with PD, 20 with PPS) who will complete 7 scheduled encounters (4 in-person visits, 3 remote visits) that occur every 3 months in an alternating manner. There will be 4 treatment groups (2 PD, 2 PPS) who will be administered intranasal bone marrow aspirate and intravenous bone marrow aspirate in a crossover pattern at three of the four in-person visits (Day 0, 6 months and 12 months).

ELIGIBILITY:
General Inclusion Criteria:

* Participants aged 40-75 years old with a diagnosis of PD or PPS (DLB, PSP, MSA, CBD with parkinsonism) based upon clinical criteria and standardized testing
* Participants time of documented PD or PPS is </= 6 years
* Participants with an anticipated survival of at least 3 years in the investigator's opinion
* Participants who are willing and able to give informed consent
* Participants who can comply with the study protocol over the 18-month duration
* Stable medical profile for 60 days prior to the initial intake screening
* Participants can ambulate at least 25m without assistance
* No known history of heparin-induced thrombocytopenia

PD Inclusion Criteria:

* Idiopathic Parkinson's disease patients who meet the MDS's Clinical Diagnostic Criteria for Parkinson's disease
* Responsive to levodopa or dopamine agonists defined by >/= 33% improvement in "Off"/"On" symptoms by MDS-UPDRS-III
* A modified Hoehn and Yahr stage of </= 3
* Neuroimaging findings are consistent with PD and absent of atrophy or other brain pathology inconsistent with PD
* "Normal" cognition as assessed by Montreal Cognitive Assessment (MoCA), with a value >/= 26

PPS Inclusion Criteria:

DLB -

* High probability of cognitive capacity to give informed consent by the Montreal Cognitive Assessment (MoCA), with a value >/= 23
* Probable DLB - DLB consortium: Two or more core clinical features are present (including features of parkinsonism for the study), or only one core clinical feature is present, but with one or more indicative biomarkers
* Core clinical features:

  * Fluctuating cognition with pronounced variations in attention and alertness
  * Recurrent visual hallucinations that are typically well-formed and detailed Rapid eye movement (REM) sleep behavior disorder (RBD), which may precede cognitive decline
* One or more spontaneous cardinal features of parkinsonism: bradykinesia, resting tremor, or rigidity
* Indicative biomarkers:

  * Reduced dopamine transporter uptake in basal ganglia demonstrated by SPECT/PET
  * Abnormal (low uptake) I-MIBG myocardial scintigraphy
  * Polysomnographic confirmation of REM sleep without atonia

PSP -

* MDS Diagnostic Criteria for probable PSP with predominant parkinsonism (PSP-P)
* Ocular motor dysfunction: vertical supranuclear gaze palsy or slow velocity of vertical saccades or frequent macro square wave jerks ("eyelid-opening apraxia")
* Ocular motor dysfunction + akinetic-rigid, axial predominant, levodopa resistant or with tremor and/or asymmetric and/or levodopa responsive (akinesia)
* "Normal" cognition as assessed by Montreal Cognitive Assessment (MoCA), with a value >/= 26

MSA -

* MDS Diagnostic Criteria for clinically probable MSA
* Autonomic dysfunction
* Parkinsonism
* Cerebellar syndrome, including at least one of gait ataxia, limb ataxia, cerebellar dysarthria, or oculomotor features
* "Normal" cognition as assessed by Montreal Cognitive Assessment (MoCA), with a value >/= 26

CBD -

* Chronic progressive course
* Asymmetric onset
* Higher cortical dysfunction: apraxia, speech apraxia, non-fluent aphasia, alien limb phenomena, or cortical sensory loss
* Movement disorder: rigid/akinetic syndrome and either dystonic limb posturing or focal myoclonus in limb, and levodopa resistant
* "Normal" cognition as assessed by Montreal Cognitive Assessment (MoCA), with a value >/= 26

Exclusion Criteria:

* Other non-PD/PPS Parkinsonism (e.g., drug-induced, vascular parkinsonism)
* No strong familial history of PD/PPS not attributable to environmental exposure or any known genetic predisposition to PD/PPS
* Unable to receive/tolerate neuroimaging (e.g., MRI-incompatible cardiac pacemaker)
* Unable to maintain/tolerate supine position with cervical neck extension
* Active systemic infection or local infection near the lumbar pelvis region
* Any bone marrow aspiration from the pelvis within 6 months of initial screening
* Any musculoskeletal-pelvis contraindications to BMA harvest from the PSIS
* Concurrent enrollment in another PD/PPS study or having taken/received another investigational intervention within 6 weeks of initial screening
* Malignancy diagnosed </= 2 years prior to initial screening
* History of intracranial or nasopharyngeal surgery deemed detrimental to the participant during the trial, including brain surgery/stereotactic procedure for PD/PPS
* History of electroconvulsive therapy
* Chronic Kidney Disorder (CKD) > Stage II or eGFR <60 mL/min
* Autoimmune disease, including:

  * Rheumatoid Arthritis (RA)
  * Systemic Lupus Erythematosus (SLE)
* Any disorders of glucocorticoid excess or diseases requiring systemic steroids or immune-modulating therapies
* Cardiac disease deemed significant:

  * Poorly controlled hypertension (BP >/=140/90)
  * NYHA class III or IV congestive heart failure
  * History of a significant ventricular arrhythmia
* Obesity class II or higher (BMI >/= 35)
* Moderate-to-uncontrolled diabetes HbA1c >/= 7%
* Osteoporosis
* A history of other severe systemic disorders, including significant CVA, TBI, seizure, encephalitis, meningitis, or psychiatric disorder that is deemed potentially harmful to the participant by the PI
* Positive for HIV, HBV, HCV, or syphilis
* Any of the following lab abnormalities:

  * Hematology: Hgb < 10 g/dl, ANC < 1.550/L, platelets < 100,000 /L >Chemistry: albumin < 3.0 g/dL, serum creatine > 1.5 x ULN, total bilirubin > 1.5 x ULN, AST/ALT/ALP > 2.0 x ULN
* Female or another gender with childbearing potential not willing to adopt barrier method(s) of contraception, plus one other form, including:

  * Intrauterine system (IUS)
  * Intrauterine device (IUD)
  * Oral, injected, or implanted hormonal contraception
* Female or another gender who is lactating/breastfeeding or has a positive urine or serum pregnancy test at intake screening
* Any disorder that compromises the participant's ability to give appropriate informed consent or hinders the ability to perform the assessment and receive the study's interventions
* Any other condition not listed above that is deemed potentially harmful to the participant by the PI

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Movement-Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS)-III | Day 0, 6, 12 and 18 months
  The MDS-UPDRS is the most widely used clinical rating scale for Parkinson disease. Part III is a motor examination (33 scores summed from 18 questions) conducted by the rater. Total scores can range from 0 to 141, with higher scores indicating worse disease severity.
10-meter Walk Test (10MWT) | Day 0, 6, 12 and 18 months
  The 10MWT is an assessment of gait speed over a short distance (2 meters ramp up, 6 meters walking, 2 meters ramp down). The aforementioned distances will be pre-measured for accuracy and only the middle 6 meters will be timed. Participants will be asked to walk at a comfortable pace for 2 trials and a fast pace for 2 trials.
Five Times Sit to Stand (FTSTS) | Day 0, 6, 12 and 18 months
  The FTSTS objectively assesses the time it takes to complete 5 sit-to-stands and is a method to observe movement strategies or compensations. The test will be performed in a standard chair with participants instructed to stand up and sit down 5 times as quickly as possible.
Mini Balance Evaluation Systems Test (Mini-BESTest) | Day 0, 6, 12 and 18 months
  The Mini-BESTest aims to target 6 different balance control systems. The measure includes 14 items assessing anticipatory postural adjustments, reactive balance control, sensory orientation, and dynamic gait. This is scored on a 3-item ordinal scale resulting in a maximum score of 28.
The Short Parkinson's Evaluation Scale (SPES)/Scales for Outcomes in Parkinson's Disease - Motor Function (SPES/SCOPA - Motor) | Day 0, 6, 12 and 18 months
  The SPES/Scales for Outcomes in Parkinson's will be used to evaluate motor function and includes 3 sections: Motor evaluation (10 items, maximum of 42 points), Activities of Daily Living (7 items, maximum 21 points), and Motor complications (4 items, maximum 12 points - with 2 items on motor fluctuation [6 points] and 2 on dyskinesias [6 points]). Response options for all items range 0 to 3.
Modified Hoehn & Yahr Scale | Day 0, 6, 12 and 18 months
  The Modified Hoehn and Yahr Scale contains additional criteria to rate Parkinson disease symptoms on a scale of 1-5. Higher scores indicate increased disease progression.
Montreal Cognitive Assessment (MoCA) | Day 0, 3, 6, 9, 12, 15 and 18 months
  The MoCA is a rapid screen of cognitive abilities to detect mild cognitive dysfunction. Participants are tested on 16 items that cover multiple cognitive domains. The score ranges from 0-30, with higher scores indicating less cognitive impairment.
Progressive Supranuclear Palsy Clinical Deficits Scale (PSP-CDS) | Day 0, 6, 12 and 18 months
  The PSP-CDS was developed to assess clinical deficits in patients with Progressive Supranuclear Palsy (PSP). The scale measures severity of deficits in seven patient-related clinical domains: Akinesia-rigidity, Bradyphrenia, Communication, Dysphagia, Eye movements, Finger dexterity, and Gait & balance; each scored from 0 to 3. The sum of the individual domains provides a total score ranging from 0 (no deficit in any domain) to 21 (severe deficit in all domains) with higher scores representing a worse outcome.
Unified Multiple System Atrophy Rating Scale (UMSARS) | Day 0, 6, 12 and 18 months
  The UMSARS will be used as a clinical rating scale to provide measures of disease progression in multiple systems atrophy. It is composed of four subscales: UMSARS-I (historical review of disease-related impairments, 12 items, scored 0 to 4), UMSARS-II (motor examination, 14 items, scored 0 to 4), UMSARS-III (autonomic examination - records blood pressure and heart rate in the supine and standing positions), and UMSARS-IV (global disability scale - rates chore-based disability, 1 item, ranges from 1 to 5). Higher scores on the UMSARS indicate greater disability.
Cortical Basal Ganglia Functional Scale (CBFS) | Day 0, 6, 12 and 18 months
  The CBFS is a rating scale that evaluates experiences in daily living (EDLs), behavioral, language, and cognitive impairments in patients with 4 repeat tauopathies (4RTs). The CBFS consists of 14 questions on Motor EDLs and 17 questions on Non-motor EDLs, each of which are rated on a Likert scale rating function from 0 to 4, where 0 = Normal or No problems and 4 = Severe problems. The questions are for the patient, but should be answered by both the patient and their caregiver together.
Parkinson's Disease Questionnaire - 39 (PDQ-39) | Day 0, 3, 6, 9, 12, 15 and 18 months
  The PDQ-39 is a self report questionnaire that assesses quality of life over the past month across 8 different dimensions (Activities of daily living, Attention and working memory, Cognition, Communication, Depression, Functional mobility, Quality of life, Social relationships, Social relationships, Social support). Items are scored based on a 5-point ordinal system with lower scores reflecting better quality of life. Each dimension total score ranges from 0 (never having difficulty) to 100 (always having difficulty) with lower scores being a better outcome.
The Scales for Outcomes in Parkinson's disease - Cognition (SCOPA-COG) | Day 0, 3, 6, 9, 12, 15 and 18 months
  The SCOPA-COG consists of 10 items divided over four domains: memory (4 items), attention (2 items), executive function (3 items), and visuospatial function (1 item). Scores range from 0-43, with higher scores reflecting better performance.
The Scales for Outcomes in Parkinson's Disease - Autonomic Dysfunction | Day 0, 3, 6, 9, 12, 15 and 18 months
  The SCOPA-AUT is self-completed by patients and consists of 23 items assessing the following domains: Gastrointestinal (7 items), Urinary (6 items), Cardiovascular (3 items), Thermoregulatory (4 items), Pupillomotor (1 item), and Sexual (2 items female, 2 items male). The maximum score is 69, with the score for each item ranging from 0 (never experiencing the symptom) to 3 (often experiencing the symptom).
Non-Motor Symptoms Questionnaire (NMSQ) | Day 0, 3, 6, 9, 12, 15 and 18 months
  The NMSQ is a comprehensive assessment of a diverse range of non-motor symptoms which can occur in all stages of Parkinson's disease. It is a patient-based screening tool designed to draw attention to the presence of non-motor symptoms in patients. Responses are marked as "yes" or "no" in regard to symptoms over the past month.
MDS Non-Motor Rating Scale (MDS-NMS) | Day 0, 3, 6, 9, 12, 15 and 18 months
  The MDS-NMS is a rater completed assessment that measures frequency and severity of 13 non-motor domains, over 52 items and covers a range of key non-motor symptoms both PD and treatment related. Scores are rated based on symptoms over the past month on frequency (scale from 0 to 4) and severity (scale 0 to 4), with higher scores reflecting more frequent and severe symptoms.

SECONDARY OUTCOMES:
Resting state brain activation pattern (fMRI analysis) | Day 0 and 18 months
  An anatomical scan using fMRI at the University of Colorado Intermountain Neuroimaging Consortium will performed during a resting state to determine changes in atrophy pattern, volume, cortical thickness, ventricle enlargement, white matter hyperintensities, and magnetic inhomogeneity effects
Active brain activation pattern (fMRI analysis) | Day 0 and 18 months
  A motor sequencing tapping task and higher order cognitive task (Stroop test) at the University of Colorado Intermountain Neuroimaging Consortium will be performed during the fMRI to determine changes in atrophy pattern, volume, cortical thickness, ventricle enlargement, white matter hyperintensities, and magnetic inhomogeneity effects.
Active performance accuracy and rate (fMRI analysis) | Day 0 and 18 months
  A motor sequencing tapping task and higher order cognitive task (Stroop test) at the University of Colorado Intermountain Neuroimaging Consortium will be performed during the fMRI to determine changes accuracy and rate of responding for motor performance and cognitive performance.

OTHER OUTCOMES:
Intranasal Bone Marrow-Mesenchymal Stem Cells (BM-MSC) Indices | Day 0, 6 and 12 months
  Number and viability of MSC's atomized
Intravenous Bone Marrow-Mesenchymal Stem Cells (BM-MSC) Indices | Day 0, 6 and 12 months
  Number and viability of MSC's infused
Bone Marrow (BM) Indices Comparative Analysis | Day 0, 6, 12 and 18 months
  Comparative analysis over the study period on the effects of multiple harvest interventions and differential cell counts on MSCs counts/viabilities
Complete Blood Count (CBC) Indices Comparative Analysis | Day 0, 6, 12 and 18 months
  Comparative analysis over the study period on the effects of multiple harvest interventions and differential cell counts on CBC counts/viabilities
Epigenetics | Day 0 and 18 months
  Analysis of DNA methylation using the DNAm Grimage, which is a linear combination of chronological age, sex, and DNAm-based surrogate biomarkers for seven plasma proteins and smoking pack-years
Metagenomics - Gut Microbiota | Day 0 and 18 months
  Stool samples will be collected from participants and sent to collaborator at Boys Town National Research Hospital to perform metagenomic shot gun sequencing and CPA/Network Analysis/MIC analysis on gut bacteria.
Metagenomics - Nasopharyngeal Microbiota | Day 0 and 18 months
  Nasopharyngeal samples will be collected from participants by a trained examiner and sent to collaborator at Boys Town National Research Hospital to perform metagenomic shot gun sequencing and CPA/Network Analysis/MIC analysis on nasopharyngeal bacteria.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Glowney, MD, MSc, Principal Investigator — Apeiron Research Center

IPD SHARING:
Plan to Share IPD: No